CLINICAL TRIAL: NCT06787651
Title: Comparison of RIMA-SVG and Ao-SVG Techniques in Coronary Artery Bypass Grafting : A Prospective Randomized Double-Blind Study on Graft Patency and Clinical Outcomes
Brief Title: Comparison of RIMA-SVG and Ao-SVG Techniques in Coronary Artery Bypass Grafting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Kexiang Liu, MD, Principal Investigator, Second Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JDEYXXGWK460
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Bypass Grafting; Coronary Artery Disease; Saphenous Vein; Graft Patency
Keywords: Coronary Artery Bypass Grafting; Saphenous Vein Graft; Graft Patency; Major Adverse Cardiovascular Events; Right Internal Mammary Artery; Neurological complications; left internal mammary artery; Surgical site infection event
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two groups based on surgical technique (RIMA-SVG vs. Ao-SVG)
Who Masked: Participant, Investigator
Masking Description: The surgical team is unblinded during the procedure, but patients and investigators remain blinded throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIMA-SVG Group (Experimental): Saphenous vein grafts (SVGs) will be connected to the right internal mammary artery (RIMA).
  Interventions: Procedure: RIMA-SVG
- Ao-SVG Group (Active Comparator): SVGs will be connected directly to the ascending aorta.
  Interventions: Procedure: Ao-SVG

INTERVENTIONS:
Procedure: RIMA-SVG — Saphenous vein grafts (SVGs) are connected to the right internal mammary artery (RIMA)
  Other Names: RIMA
  Arms: RIMA-SVG Group
Procedure: Ao-SVG — The ascending aorta is clamped, and SVGs are anastomosed to the aorta.
  Other Names: Ao
  Arms: Ao-SVG Group

SUMMARY:
This randomized, double-blind, single-center clinical trial was divided into two groups, RIMA-SVG and Ao-SVG, according to the surgical method. The purpose was to evaluate the effect of the RIMA-SVG surgical method in improving saphenous vein graft (SVG) patency and reducing clinical complications. A total of 300 patients will be enrolled and randomly assigned to two surgical method groups: RIMA-SVG Group (150 patients): SVGs are connected to the right internal mammary artery (RIMA). Ao-SVG Group (150 patients): The aorta is clamped, and SVGs are connected to the ascending aorta (Ao).All patients will undergo CABG on a beating heart with sequential vein grafts to bypass at least two or more coronary vessels. The primary outcome is 1-year graft patency. The secondary outcomes include neurological complications, mortality, major adverse cardiovascular events (MACE), and surgical site infection event.

DETAILED DESCRIPTION:
This randomized, double-blind, single-center clinical trial was divided into two groups, RIMA-SVG and Ao-SVG, according to the surgical method. The purpose was to evaluate the effect of the RIMA-SVG surgical method in improving saphenous vein graft (SVG) patency and reducing clinical complications. A total of 300 patients undergoing CABG on a beating heart will be randomized into two surgical technique groups: RIMA-SV Group (150 patients): SVGs are anastomosed to the right internal mammary artery (RIMA). Ao-SVG Group (150 patients): The ascending aorta is clamped, and SVGs are anastomosed to the aorta. All patients will undergo CABG via median sternotomy, and the left internal mammary artery (LIMA) will be used to bypass the left anterior descending artery (LAD). SVGs will be sequentially grafted to the circumflex artery, diagonal branch, and right coronary artery. The primary outcome is 1-year graft patency, assessed by coronary CT angiography and classified using the FitzGibbon grading system. Secondary outcomes include all-cause mortality, major adverse cardiovascular events (MACE), neurological complications, and surgical site infection event. Patients will be followed at 12 months for clinical evaluations and imaging assessments. Inclusion criteria include patients aged 18 to 80 years undergoing planned CABG with at least two sequential saphenous vein grafts and who are able to provide written informed consent. Exclusion criteria include additional cardiac surgeries, severe subclavian artery stenosis, unsuitable SVGs (e.g. bilateral varicosities), history of intracranial hemorrhage, active bleeding, malignancy, or emergency surgery. Randomization will be computer-generated, and all aspects of the study will remain blinded to ensure unbiased assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years.
2. Scheduled for their first planned coronary artery bypass grafting (CABG) with at least two sequential saphenous vein grafts (SVGs).
3. Able and willing to provide written informed consent.

Exclusion Criteria:

1. Patients unable to provide written informed consent.
2. Patients requiring other cardiac surgeries (e.g. valve replacement, congenital heart defect surgery, or aortic dissection repair).
3. Patients with severe stenosis of the left or right subclavian artery.
4. Patients for whom aortic clamping is infeasible due to calcification of the ascending aorta.
5. Patients with bilateral SVG varicosities unsuitable for grafting.
6. Patients with active malignancy.
7. Patients with active bleeding or a history of bleeding tendency.
8. Patients with previous intracranial hemorrhage, ischemic stroke within 14 days preoperatively, or severe carotid artery stenosis.
9. Patients with severe hepatic dysfunction.
10. Patients requiring emergency surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
1-Year Graft Patency | 1 year post-surgery
  The patency of saphenous vein grafts (SVGs) will be assessed 1 year post-surgery using coronary CT angiography

SECONDARY OUTCOMES:
Perioperative complications | 2 weeks post-surgery
  Incidence of Perioperative complications related to CABG, including myocardial infarction, arrhythmias and other major adverse events.
Neurological Complications | 1 year post-surgery
  Incidence of neurological complications, including stroke within 1 year after CABG.
All-Cause Mortality | 1 year post-surgery
  Incidence of MACCE, including cardiovascular death, non-fatal myocardial infarction, Incidence of death from any cause within 1 year after CABG.
Major Adverse Cardiovascular Events (MACE) | 1 year post-surgery
  Incidence of MACCE, including cardiovascular death, non-fatal myocardial infarction, and target vessel revascularization, within 1 year after CABG.after CABG.
Surgical site infection event | 1 year post-surgery
  Incidence of surgical site infection event during hospitalization and within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: kexiang liu, Ph.D., Study Director — Second Hospital of Jilin University
Locations (1):
- the Second Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcomes of the study-including baseline characteristics, graft patency results, perioperative complications, and 12-month clinical outcomes-will be made available upon reasonable request. Data will be shared with qualified researchers following study completion and publication, subject to approval by the trial steering committee and in accordance with ethical and data protection guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be shared via request from the corresponding author starting 6 months after study completion and publication.
Access Criteria: Access to the de-identified individual participant data will be granted to qualified researchers whose proposed use of the data has been reviewed and approved by the trial's principal investigator and data access committee. Applicants must submit a detailed research proposal outlining the scientific rationale, intended analyses, and data protection measures. A data use agreement must be signed prior to data release to ensure compliance with ethical and legal standards.

REFERENCES:
- [Derived] Wei R, Huang M, Jiang N, Zhang R, He T, Zhu C, Wang W, Piao H, Yu S, Zhu Z, Wang T, Liu K. RIMA-SVG versus Ao-SVG in coronary artery bypass grafting: protocol for a prospective, randomised, double-blind, non-inferiority and single-centre trial. BMJ Open. 2025 Sep 28;15(9):e104578. doi: 10.1136/bmjopen-2025-104578. PMID 41022447